CLINICAL TRIAL: NCT02240797
Title: Kappa Opioid Receptor Imaging in Anorexia
Status: Terminated | Type: Observational
Why Stopped: The original PI, Alexander Neumeister, left NYULMC. No data was analyzed.
Sponsor: NYU Langone Health (Other)
Collaborators: Yale University (Other); Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Other Study IDs: S13-00990
Record Dates: First submitted 2014-09-09; First posted 2014-09-16 (Estimated); Last update posted 2016-08-17 (Estimated); Status verified 2016-08

CONDITIONS: Anorexia Nervosa
Keywords: Anorexia Nervosa; Neuroimaging; Positron emission tomography (PET); [11C]PKAB
MeSH Terms: conditions — Anorexia Nervosa | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Anorexia Nervosa - Recovered (AN-REC): Anorexia Nervosa - Recovered (AN-REC)
  Interventions: Other: Positron emission tomography (PET) imaging
- Healthy Control (HC): Healthy Control (HC)
  Interventions: Other: Positron emission tomography (PET) imaging

INTERVENTIONS:
Other: Positron emission tomography (PET) imaging — Positron emission tomography (PET) imaging

SUMMARY:
The purpose of this study is to use positron emission tomography (PET) imaging and magnetic resonance imaging (MRI) to understand the brain function of individuals with anorexia nervosa and healthy controls.

DETAILED DESCRIPTION:
This is a 3-year study involving n=7 women with anorexia nervosa - recovered (AN-REC) from restricting subtype that have achieved a body mass index (BMI) > 18.5 in the past year, are medication free, range in age from 18-55 years and n=7 healthy (medical and psychiatric statues) age- and weight-matched controls who are invited to participate in a medical and psychiatric evaluation, neuroendocrine assessments, one magnetic resonance imaging (MRI) study and one positron emission tomography (PET) study kappa opioid receptor (KOR) 11-carbon (11C) [11C]PKAB and PET. Subjects will be asked to provide written informed consent after full explanation of all study procedures and risks and benefits related to study participation. On the screening day a full medical evaluation including blood work, urine analyses, toxicology, electrocardiogram (ECG) and physical exam will be performed.

ELIGIBILITY:
Inclusion criteria for anorexic patients:

1. Able to understand the consent form document
2. A willingness to participate in a psychiatric evaluation, collection of behavioral ratings and neuroendocrine assessments, and imaging studies including 1 PET scan and 1 MRI scan
3. Meets criteria for Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) Anorexia Nervosa (AN)
4. Subjects will be between 18 and 55 years of age
5. Currently weight restored with a body mass index (BMI) > 18.5 for longer than 3 months

Inclusion criteria for healthy controls:

1. Able to understand the consent form document
2. A willingness to participate in a psychiatric evaluation, collection of behavioral ratings and neuroendocrine assessments, and imaging studies including 1 PET scan and 1 MRI scan
3. Subjects will be between 18 and 55 years of age
4. Regular menstruation and no personal or first-degree family history of any Axis I diagnosis based on DSM-IV criteria

Exclusion criteria for anorexic patients:

1. Any major neurological illness or injury
2. Presence of any legal or illegal psychoactive substances determined with urine toxicology, and breathalyzer test for alcohol
3. Any significant unstable medical condition such as asthma or heart disease which may limit the interpretation of the imaging results, for example due to changes in tracer delivery in hypertensive patients
4. Intelligence quotient (IQ)<70 based on past intelligence
5. Any metal in body that would pose a risk with MRI
6. Claustrophobia that would interfere with MRI or PET imaging
7. Currently pregnant or nursing

Exclusion criteria for healthy controls:

1. Any major neurological illness or injury
2. Presence of any legal or illegal psychoactive substances determined with urine toxicology, and breathalyzer test for alcohol
3. Any significant unstable medical condition such as asthma or heart disease which may limit the interpretation of the imaging results, for example due to changes in tracer delivery in hypertensive patients
4. IQ<70 based on past intelligence
5. Any metal in body that would pose a risk with MRI
6. Claustrophobia that would interfere with MRI or PET imaging
7. Currently pregnant or nursing

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Subjects are female, between the age range of 18 to 55, are medically healthy and currently not taking any medications to treat any medical illness, and have a history of anorexia nervosa and are recovered or never had a history of anorexia nervosa.
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2014-09; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Volume of distribution (VT) (i.e., KOR binding) using [11C]PKAB and PET imaging | Two months
  In this study we are using the KOR radioligand [11C]PKAB and PET to investigate group differences in cerebral KOR binding potential in 7 AN-REC and 7 healthy controls (HCs).

CONTACTS AND LOCATIONS:
Overall Officials: Charles Marmar, MD, Principal Investigator — NYU School of Medicine
Locations (1):
- NYU School of Medicine, New York, New York, United States